CLINICAL TRIAL: NCT00021125
Title: A Randomized Controlled Trial Of CHARTWEL (a Continuous Hyperfractionated Accelerated Radiotherapy Schedule) Versus Conventional Radiotherapy In Post-Operative Head And Neck Cancer Patients
Brief Title: Radiation Therapy in Treating Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MRC-CH03; CDR0000068750 (Registry Identifier: PDQ (Physician Data Query)); EU-20121; ISRCTN62576956
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2002-12

CONDITIONS: Head and Neck Cancer; Non-melanomatous Skin Cancer
Keywords: squamous cell carcinoma of the skin; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known which regimen of radiation therapy is more effective for head and neck cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of different regimens of radiation therapy in treating patients who have head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare adjuvant continuous hyperfractionated accelerated radiotherapy vs conventional radiotherapy, in terms of preventing disease recurrence, in patients with head and neck cancer.
* Compare the early and late toxic effects of these treatments in this patient population.
* Compare disease-free and overall survival of patients receiving these treatments.
* Assess quality of life in patients receiving these treatments.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms.

* Arm I: Patients undergo radiotherapy 3 times daily, with an interval of at least 6 hours between any 2 treatments, 5 days a week, for just over 2 weeks, for a total of 13-14 treatment days.
* Arm II: Patients undergo radiotherapy daily, 5 days a week, for 6-6.5 weeks. Quality of life is assessed at baseline and then annually for 5 years.

Patients are followed every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 460 patients (230 per arm) will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck including, but not limited to, the following:

  * Oral cavity
  * Oropharynx
  * Hypopharynx
  * Larynx
  * Nasal sinuses
  * Skin
* Undergone curative surgery within the past 70 days

  * All macroscopic disease removed
* At high or intermediate risk of recurrence

  * No low risk of recurrence
* No evidence of distant metastases
* Considered treatable by radiotherapy

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other prior or concurrent malignancy that would preclude study participation
* No other uncontrolled medical illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2000-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Time to local recurrence

SECONDARY OUTCOMES:
Length of survival
Morbidity and toxicity
Quality of life as assessed by EORTC Quality of life Questionnaire for Head and Neck Cancer

CONTACTS AND LOCATIONS:
Overall Officials: M. I. Saunders, MD, Study Chair — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (1):
- Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England, United Kingdom